CLINICAL TRIAL: NCT03149094
Title: Feasibility and Acceptability of an mHealth Cognitive Behavioral Stress Management Intervention to Ameliorate HIV-related Fatigue
Brief Title: CBSM Intervention Via mHealth to Ameliorate HIV-related Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00057504; 1P20NR016575-01 (NIH)
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: HIV; Stress Disorder; Human Immunodeficiency Virus; Fatigue
Keywords: Self-Management; mHealth
MeSH Terms: conditions — Stress Disorders, Traumatic; Acquired Immunodeficiency Syndrome; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBSM-SMI (Experimental): The intervention group will receive Cognitive Behavioral Stress Management (CBSM) for Individuals Living with HIV via mHealth through smartphones and tablets.
  Interventions: Behavioral: CBSM-SMI
- CBSM-SMI control (Active Comparator): The control group will receive an app called LifeSum, which focuses on healthy lifestyles.
  Interventions: Behavioral: CBSM-SMI control

INTERVENTIONS:
Behavioral: CBSM-SMI — The intervention group will receive Cognitive Behavioral Stress Management (CBSM) for Individuals Living with HIV via mHealth through smartphones and tablets.
  Arms: CBSM-SMI
Behavioral: CBSM-SMI control — this group will receive the LifeSum app.
  Arms: CBSM-SMI control

SUMMARY:
The purpose of this study is to create a smartphone, tablet and web-based application to help people deal with stress. Stress often increases fatigue in people with HIV infection, so successfully dealing with stress could help reduce HIV-related fatigue. The study is being done at one site, the Medical University of South Carolina. Approximately 30 people will take part in this portion of the study.

DETAILED DESCRIPTION:
For this study we will develop a fatigue symptom self-management cognitive behavioral stress management (CBSM) program that will be delivered via mHealth through smartphones and tablets (optimized for each). All CBSM content will be integrated into the application, but tailoring of information delivery will be derived through algorithm-driven feedback based on user input as they respond to integrated assessment and symptom monitoring questions. As a result, users of the CBSM-Self Management Intervention (CBSM-SMI) will receive personalized, relevant intervention content, when they need it, where they need it. This novel mode of CBSM delivery has not yet been provided via an mHealth format to HIV-infected individuals, despite its obvious advantages insofar as cost and reach are concerned.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Reads and understands English
* Scores greater than 5 on the HIV-Related Fatigue Scale
* Mentally competent to give informed consent

Exclusion Criteria:

* Co-morbid conditions marked by fatigue (e.g., renal disease, cancer, multiple sclerosis)
* Pregnant women and women who are less than 1 year postpartum
* Active psychosis or dementia
* Suicidal ideation with clear intent
* Current substance dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability Scale | Baseline
  The Feasibility and Acceptability Scale is a 5 item, 5-point scale, developed to assess the feasibility and acceptability of interventions.
Feasibility and Acceptability Scale | 10 weeks
  The Feasibility and Acceptability Scale is a 5 item, 5-point scale, developed to assess the feasibility and acceptability of interventions.
Feasibility and Acceptability Scale | 22 weeks
  The Feasibility and Acceptability Scale is a 5 item, 5-point scale, developed to assess the feasibility and acceptability of interventions.

SECONDARY OUTCOMES:
HIV-Related Fatigue Scale (HRFS) | Baseline
  The HRFS is a 56-item instrument which assesses fatigue severity, responsiveness to self-care, and fatigue-related impairment of functioning in HIV infection.
HIV-Related Fatigue Scale (HRFS) | 5 weeks
  The HRFS is a 56-item instrument which assesses fatigue severity, responsiveness to self-care, and fatigue-related impairment of functioning in HIV infection.
HIV-Related Fatigue Scale (HRFS) | 10 weeks
  The HRFS is a 56-item instrument which assesses fatigue severity, responsiveness to self-care, and fatigue-related impairment of functioning in HIV infection.
HIV-Related Fatigue Scale (HRFS) | 22 weeks
  The HRFS is a 56-item instrument which assesses fatigue severity, responsiveness to self-care, and fatigue-related impairment of functioning in HIV infection.
PROMIS Short Form - Fatigue 8a | Baseline
  The PROMIS Fatigue 8a evaluates a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social role.
PROMIS Short Form - Fatigue 8a | 5 weeks
  The PROMIS Fatigue 8a evaluates a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social role.
PROMIS Short Form - Fatigue 8a | 10 weeks
  The PROMIS Fatigue 8a evaluates a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social role.
PROMIS Short Form - Fatigue 8a | 22 weeks
  The PROMIS Fatigue 8a evaluates a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social role.
The State Trait Anxiety Inventory (STAI)-State | Baseline
  The STAI is a self-report measure of state anxiety, consisting of 20 emotion descriptor items; respondents indicate how they are feeling right now by rating each item on a 4-point scale.
The State Trait Anxiety Inventory (STAI)-State | 5 weeks
  The STAI is a self-report measure of state anxiety, consisting of 20 emotion descriptor items; respondents indicate how they are feeling right now by rating each item on a 4-point scale.
The State Trait Anxiety Inventory (STAI)-State | 10 weeks
  The STAI is a self-report measure of state anxiety, consisting of 20 emotion descriptor items; respondents indicate how they are feeling right now by rating each item on a 4-point scale.
The State Trait Anxiety Inventory (STAI)-State | 22 weeks
  The STAI is a self-report measure of state anxiety, consisting of 20 emotion descriptor items; respondents indicate how they are feeling right now by rating each item on a 4-point scale.
Beck Depression Inventory (BDI-II) | Baseline
  The BDI-II is a 21 item measure of depressive severity with higher total scores indicative of more severe depression.
Beck Depression Inventory (BDI-II) | 5 weeks
  The BDI-II is a 21 item measure of depressive severity with higher total scores indicative of more severe depression.
Beck Depression Inventory (BDI-II) | 10 weeks
  The BDI-II is a 21 item measure of depressive severity with higher total scores indicative of more severe depression.
Beck Depression Inventory (BDI-II) | 22 weeks
  The BDI-II is a 21 item measure of depressive severity with higher total scores indicative of more severe depression.
Life Experiences Scale | Baseline
  The Life Experiences Scale is a 30-item self-report measure that allows respondents to indicate recent stressful life events.
Life Experiences Scale | 5 weeks
  The Life Experiences Scale is a 30-item self-report measure that allows respondents to indicate recent stressful life events.
Life Experiences Scale | 10 weeks
  The Life Experiences Scale is a 30-item self-report measure that allows respondents to indicate recent stressful life events.
Life Experiences Scale | 22 weeks
  The Life Experiences Scale is a 30-item self-report measure that allows respondents to indicate recent stressful life events.
CD4 count from the medical record | Baseline
  A CD4 count is a lab test that measures the number of CD4 T lymphocytes (CD4 cells) in a sample of blood. In people with HIV, it is the most important laboratory indicator of how well the immune system is working and the strongest predictor of HIV progression.
CD4 count from the medical record | 22 weeks
  A CD4 count is a lab test that measures the number of CD4 T lymphocytes (CD4 cells) in a sample of blood. In people with HIV, it is the most important laboratory indicator of how well the immune system is working and the strongest predictor of HIV progression.
HIV viral load information from the medical record | Baseline
  A viral load test is a lab test that measures the number of HIV virus particles in a milliliter of blood. A viral load test helps provide information on how well antiretroviral therapy is controlling the virus.
HIV viral load information from the medical record | 22 weeks
  A viral load test is a lab test that measures the number of HIV virus particles in a milliliter of blood. A viral load test helps provide information on how well antiretroviral therapy is controlling the virus.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barroso J, Madisetti M, Mueller M. A Feasibility Study to Develop and Test a Cognitive Behavioral Stress Management Mobile Health Application for HIV-Related Fatigue. J Pain Symptom Manage. 2020 Feb;59(2):242-253. doi: 10.1016/j.jpainsymman.2019.09.009. Epub 2019 Sep 17. PMID 31539601